CLINICAL TRIAL: NCT01118845
Title: A Multinational, Multicenter, Open-Label Phase II Study of SyB L-0501 in Combination With Rituximab in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Study of SyB L-0501 in Combination With Rituximab to Treat Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Masahiro Furukawa, SymBio Pharmaceuticals Limited
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010001
Record Dates: First submitted 2010-05-01; First posted 2010-05-07 (Estimated); Results first posted 2013-07-04 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-05

CONDITIONS: Non-Hodgkin's Lymphoma; Lymphoma, Large Cell; Diffuse, Mantle Cell Lymphoma, Lymphoma; Follicular Lymphoma; Large B-Cell, Diffuse
Keywords: Non-Hodgkin's lymphoma; Lymphoma, Large B-Cell; Diffuse, Mantle cell lymphoma, Lymphoma; Follicular, Lymphoma; Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma; Lymphoma, Follicular | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SyB L-0501 (Experimental)
  Interventions: Drug: SyB L-0501; Drug: Rituximab

INTERVENTIONS:
Drug: SyB L-0501 — The administration of SyB L-0501 at 120 mg/m^2/day by intravenous infusion on day 2 and 3 of each 21-day cycle with up to 6 cycles. Dose modifications are permitted from 2nd cycle according to dose reduction schedule.
  SyB L-0501 60 mg/m^2, 90 mg/m^2 or 120 mg/m^2/day on Day 2 and Day 3 will be followed by 18 days of observation.
  Other Names: Bendamustine hydrochloride
Drug: Rituximab — The administration of rituximab at 375 mg/m^2/day by intravenous infusion on day 1 of each 21-day cycle with up to 6 cycles. Dose modifications are not permitted.

SUMMARY:
The purpose of this study is to determine the efficacy of SyB L-0501 in combination with rituximab in patients with relapsed/refractory diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
Primary Objective is to determine the efficacy, as measured by overall response rate on the basis of Revised Response Criteria for Malignant Lymphoma, of SyB L-0501 at 120 mg/m^2/day on day2 and 3 in combination with rituximab at 375 mg/m^2 on day 1 of each 21-day cycle in patients with relapsed/refractory diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented Cluster of differentiation 20 (CD20)-positive for lymphoma cells
* Patients with measurable lesions
* Patients with measurable lesions >1.5 cm in major axes
* Relapsed or refractory after 1 to 3 prior therapeutic treatments for diffuse large B-cell lymphoma.
* Patients who are expected to survive for at least 3 months
* Patients aged from 20 to 75 years at the time informed consent is obtained
* Performance Status (P.S.) of 0 to 1 at initial administration of the study drug
* Patients with adequately maintained organ functions
* Patients capable of personally giving voluntary informed consent in writing to participate in the study

Exclusion Criteria:

* Patients who have been without treatment for less than 3 weeks after prior treatment
* Patients who can be candidates for autologous peripheral blood stem cell transplantation at the discretion of the investigator.
* Patients who received adequate prior treatments and did not respond to any of them.
* Patients with central nervous system (CNS) involvement or patients with clinical symptoms suggestive of CNS involvement.
* Patients with serious, active infections
* Patients with serious complications
* Patients with complications or medical history of serious cardiac disease
* Patients with serious gastrointestinal symptoms
* Patients with malignant pleural effusion, cardiac effusion, or ascites retention
* Patients positive for hepatitis B surface (HBs) antigen, hepatitis C virus (HCV) antibody, or HIV antibody
* Patients with serious bleeding tendencies
* Patients with a fever of 38.0°C or higher
* Patients with, or confirmed in the past to have had, interstitial pneumonia, pulmonary fibrosis, or pulmonary emphysema
* Patients with active multiple primary cancer or patients with a history of other malignant cancer within the past 5 years, except for basal cell cancer of the skin, squamous cell cancer, or cervical cancer in situ
* Patients with, or confirmed in the past to have had, autoimmune hemolytic anemia
* Patients who received SyB L-0501 in the past
* Patients who received cytokine preparation such as erythropoietin or granulocyte colony-stimulating factor (G-CSF) or blood transfusions within 2 weeks before the examination at registration for this study
* Patients who received other investigational products or unapproved medication within 3 months before registration in this study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kensei Tobinai, MD, Ph D, Study Chair — National Cancer Center Hospital
Locations (25):
- Japan (18):
  - Nagoya, Aichi-ken
  - Akita, Akita
  - Matsuyama, Ehime
  - Fukuoka, Fukuoka
  - Kurume, Fukuoka
  - Maebashi, Gunma
  - Sapporo, Hokkaido
  - Kanazawa, Ishikawa-ken
  - Kagoshima, Kagoshima-ken
  - Isehara, Kanagawa
  - Ninomaru, Kumamoto
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Kita-ku, Okayama-ken
  - Kurashiki, Okayama-ken
  - Hidaka, Saitama
  - Izumo, Shimane
  - Chuo-ku, Tokyo
- South Korea (7):
  - Seo-gu, Busan
  - Jung-gu, Daegu
  - Goyang-si, Gyeonggi-do
  - Hwasun-gun, Jeollanam-do
  - Gangnam-gu, Seoul
  - Seodaemun-gu, Seoul
  - Songpa-gu, Seoul

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Among the 63 subjects enrolled in the study, 59 subjects received study drug and four subjects were excluded before the first study drug administration. The reasons for exclusion were adverse events and major protocol deviation/violation for two subjects each.
Groups:
- SyB L-0501: SyB L-0501 was administered in combination with rituximab. SyB L-0501 was administered at 120 mg/m^2/day by intravenous infusion on day 2 and 3 of each 21-day cycle with up to 6 cycles. Dose modifications are permitted from 2nd cycle according to dose reduction schedule. Rituximab was administered at 375 mg/m^2/day by intravenous infusion on day 1 of each 21-day cycle with up to 6 cycles. Dose modifications are not permitted.
Period: Overall Study
Arm/Group | SyB L-0501
Started | 59
Completed | 17
Not Completed | 42

BASELINE CHARACTERISTICS:
Arm/Group | SyB L-0501
Number analyzed (Participants) | 59
Age Continuous [Mean (Standard Deviation); unit: Year] | 64.2 (9.2)
Age, Customized [Number; unit: Percentage of participants]
  20-29 years | 0.0
  30-39 years | 1.7
  40-49 years | 8.5
  50-59 years | 16.9
  60-69 years | 39.0
  70-75 years | 33.9
Age, Customized [Number; unit: Percentage of participants]
  <65 years | 37.3
  ≥65 years | 62.7
Sex/Gender, Customized [Number; unit: percentage of participants]
  Male | 42.4
  Female | 57.6
Diagnosis of Relapsed/Refractory Diffuse Large B-Cell Lymphoma [Number; unit: percentage of participants] | 100.0
Clinical Stage (Ann Arbor staging) [Number; unit: Percentage of participants] — The criteria for Clinical Stage (Ann Arbor staging) are as below:
  I: involvement of a single nodal region. II: involvement of 2 or more lymph node regions on the same side of the diaphragm. III: involvement of lymph node regions on both sides of the diaphragm. IV: disseminated involvement of 1 or more extra-lymphatic sites with or without associated lymph node involvement
  E: if accompanied by localized involvement of a extra-lymphatic organ or site. S: if accompanied by involvement of the spleen. SE: if both S and E
  Percentage of participants
    Stage I | 5.1
    Stage I-E | 3.4
    Stage II | 27.1
    Stage II-E | 3.4
    Stage III | 25.4
    Stage III-S | 6.8
    Stage III-E | 3.4
    Stage III-SE | 0.0
    Stage IV | 25.4
    Unknown | 0.0
Systemic symptoms (B symptoms) (Ann Arbor staging) [Number; unit: Percentage of participants]
  Asymptomatic | 86.4
  Symptomatic | 13.6
  Unknown | 0.0
Medical history of diffuse large B-cell lymphoma (DLBCL) [Number; unit: Percentage of participants]
  No | 40.7
  Yes | 59.3
Complications of DLBCL [Number; unit: Percentage of participants]
  No | 6.8
  Yes | 93.2
Prior medication/therapy for DLBCL [Number; unit: Percentage of participants]
  No | 8.5
  Yes | 91.5
Prior medication/therapy for DLBCL (Transplant) [Number; unit: Percentage of participants]
  No | 86.4
  Yes | 13.6
Prior treatment for DLBCL [Number; unit: Percentage of participants]
  No | 0.0
  Yes | 100.0
Number of regimens [Number; unit: Percentage of participants]
  1 | 64.4
  2 | 22.0
  3 | 13.6
P.S.(performance status)[the Eastern Cooperative Oncology Group (ECOG) criteria] [Number; unit: Percentage of Participants] — P.S.(ECOG) criteria are as below:
  0: Fully active, able to carry on all pre-disease performance without restriction. 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. 2: Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours. 3: Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours. 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  Percentage of Participants
    0 | 66.1
    1 | 33.9
Tumor diameter [Number; unit: Percentage of Participants]
  <5 cm | 71.2
  ≥5 cm | 28.8
Tumor diameter [Number; unit: Percentage of Participants]
  <7 cm | 86.4
  ≥7 cm | 13.6
lactate dehydrogenase (LDH) [Number; unit: Percentage of Participants] — The normal ranges vary among institutions.
  Percentage of Participants
    Within normal range | 44.1
    Elevated | 55.9
LDH [Number; unit: Percentage of Participants]
  <240 IU/L | 39.0
  ≥240 IU/L | 61.0
Site of disease [Number; unit: Percentage of Participants]
  <4 nodular sites | 47.5
  ≥4 nodular sites | 52.5
Site of disease [Number; unit: Percentage of Participants]
  <2 extranodular sites | 93.2
  ≥4 extranodular sites | 6.8
Bone marrow involvement [Number; unit: Percentage of Participants]
  Positive | 3.4
  Negative | 94.9
  Indeterminate | 0.0
  Unknown | 1.7
Response to prior treatment [Number; unit: Percentage of Participants]
  Responder | 100.0
  Non-Responder | 0.0
  Unknown | 0.0
Time from prior treatment [Number; unit: Percentage of Participants] — Time from the initiation of prior treatment to the initiation of the study drug in subjects with 1 regimen of prior treatment (64.4% of all the subjects).
  Percentage of Participants
    <12 months | 15.3
    ≥12 months | 49.2
    Unknown | 0.0
International Prognostic Index risk category [Number; unit: Percentage of Participants] — The criteria for International Prognostic Index risk category are as below:
  Low (score=0-1): 5-year survival of 73%. Low (score=2): 5-year survival of 51%. High-intermediate (score=3): 5-year survival of 43%. High (score=4-5): 5-year survival of 26%
  Percentage of Participants
    Low (score=0-1) | 33.9
    Low-Intermediate (score=2) | 35.6
    High-Intermediate (score=3) | 23.6
    High(score=4-5) | 6.8
    Unknown | 0.0
International Prognostic Index risk category [Number; unit: Percentage of Participants]
  Low-Intermediate (score<3) | 69.5
  High-Intermediate (score≥3) | 30.5
  Unknown | 0.0
Height [Mean (Standard Deviation); unit: cm] | 158.25 (8.59)
Weight [Mean (Standard Deviation); unit: kg] | 57.64 (12.85)
Body Surface Area（BSA） [Mean (Standard Deviation); unit: m^2] | 1.537 (0.184)

OUTCOME MEASURES:

1. Primary Outcome: The Overall Response Rate [Complete Response (CR) + Partial Response (PR)] Determined on the Basis of Revised Response Criteria for Malignant Lymphoma
Description: CR: Disappearance of all evidence of disease. PR: Regression of measurable disease and no new sites.
  For the criteria for CR, See Outcome measure 2 description.
  The criteria for PR is as below.
  Nodal Masses:
  more than 50% decrease in sum of the product of the perpendicular diameters (SPD) of up to 6 largest dominant masses; no increase in size of other nodes
  1. FDG-avid or PET positive prior to therapy; one or more PET positive at previously involved site
  2. Variably FDG-avid or PET negative; regression on CT
  Spleen, Liver:
  more than 50% decrease in SPD of nodules (for single nodule in greatest transverse diameter); no increase in size of liver or spleen
  Bone Marrow:
  Irrelevant if positive prior to therapy; cell type should be specified
Time Frame: up to 30 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 59
Percentage of Participants | 62.7 [49.1 to 75.0]

2. Secondary Outcome: The Complete Response (CR) Rate Determined on the Basis of Revised Response Criteria for Malignant Lymphoma
Description: The criteria for CR is as below
  Nodal Masses:
  1. fluorodeoxy glucose (FDG)-avid or positron emission tomography (PET) positive prior to therapy; mass of any size permitted if PET negative
  2. Variably FDG-avid or PET negative; regression to normal size on computed tomography (CT)
  Spleen, Liver:
  Not palpable, nodules disappeared
  Bone Marrow:
  Infiltrate cleared on repeat biopsy; if indeterminate by morphology, immunohistochemistry should be negative
Time Frame: up to 30 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 59
Percentage of participants | 37.3 [25.0 to 50.9]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS = day of the first PFS event - day of start of study treatment + 1
  The definitions of PFS event are as below.
  1. PD according to overall response on the basis of Revised Response Criteria for Malignant Lymphoma
     PD: Any new lesion or increase by ≥50% of previously involved sites from nadir. Nodal masses; Appearance of a new lesion(s) >1.5 cm in any axis, ≥50% increase in SPD of more than one node, or ≥50% increase in longest diameter of a previously identified node >1 cm in short axis. Lesions PET positive if FDG-avid lymphoma or PET positive prior to therapy. Spleen, Liver; ≥50% increase from nadir in the SPD of any previous lesions. Bone marrow; New or recurrent involvement
  2. Disease progression during treatment period
  3. Disease progression during follow up period
  4. Start of treatment of new lesion
  5. Occurrence of other multiple malignant tumors
  6. Death
Time Frame: up to 30 weeks
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | SyB L-0501
Number analyzed (Participants) | 59
Days | 200.0 [109.0 to 410.0]

4. Secondary Outcome: Number of Subjects With Adverse Event
Time Frame: up to 30 weeks
Measure: Number; unit: Participants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 59
Participants
  Subjects with adverse event | 59
  Subjects with serious adverse event | 14

5. Secondary Outcome: Number of Adverse Events
Time Frame: up to 30 weeks
Measure: Number; unit: Events
Arm/Group | SyB L-0501
Number analyzed (Participants) | 59
Events
  Adverse events | 1848
  Serious adverse events | 23

6. Secondary Outcome: Number of Subjects With Abnormality (Grade ≥3) in Laboratory Test Values
Description: Abnormalities in laboratory test values in overall study period were analyzed. Severity of abnormalities were evaluated using Common Terminology Criteria for Adverse Events (CTCAE).
  grade 1 : mild grade 2 : moderate grade 3 : severe grade 4 : life threatening or disabling grade 5 : death related to adverse event
Time Frame: up to 30 weeks
Measure: Number; unit: Participants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 59
Participants
  Subjects with grade 3 abnormality | 2
  Subjects with grade 4 abnormality | 54

7. Secondary Outcome: Number of Subjects With Grade ≥3 Physical Examination Finding
Time Frame: up to 30 weeks
Measure: Number; unit: Participants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 59
Participants
  Subjects with grade 3 Physical Findings | 1
  Subjects with grade 4 Physical Findings | 22

8. Secondary Outcome: Concomitant Medication Usage
Time Frame: up to 30 weeks
Measure: Number; unit: Participants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 59
Participants
  concomitant medications for adverse events | 58
  concomitant medications for complications | 50
  concomitant medications for supportive therapy | 59
  concomitant medications for other reasons | 59

9. Secondary Outcome: The Maximum Concentration (Cmax) of Unchanged SyB L-0501 in Japan
Time Frame: Prior to and 30 min after start of administration, and 0, 30, 60, 120 min after completion of administration on Day 2 of the 1st cycle
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SyB L-0501
Number analyzed (Participants) | 10
ng/mL | 8365.82 (3522.73)

10. Secondary Outcome: The Maximum Drug Concentration Time (Tmax) of Unchanged SyB L-0501 in Japan
Time Frame: as for outcome 9
Measure: Median (Standard Deviation); unit: hour
Arm/Group | SyB L-0501
Number analyzed (Participants) | 10
hour | 1.0 (0.0)

11. Secondary Outcome: The Area Under the Curve (AUC) for Unchanged SyB L-0501 in Japan
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng・h/mL
Arm/Group | SyB L-0501
Number analyzed (Participants) | 10
ng・h/mL | 10394.39 (5368.77)

12. Secondary Outcome: The Half-life Period (t1/2) of Unchanged SyB L-0501 in Japan
Time Frame: as for outcome 9
Measure: Median (Standard Deviation); unit: hour
Arm/Group | SyB L-0501
Number analyzed (Participants) | 10
hour | 0.39 (0.1)

13. Secondary Outcome: The Maximum Concentration (Cmax) of Unchanged SyB L-0501 in Korea
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SyB L-0501
Number analyzed (Participants) | 4
ng/mL | 8095.99 (4339.74)

14. Secondary Outcome: The Maximum Drug Concentration Time (Tmax) of Unchanged SyB L-0501 in Korea
Time Frame: as for outcome 9
Measure: Median (Standard Deviation); unit: hour
Arm/Group | SyB L-0501
Number analyzed (Participants) | 4
hour | 0.9 (0.3)

15. Secondary Outcome: The Area Under the Curve (AUC) for Unchanged SyB L-0501 in Korea
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng・h/mL
Arm/Group | SyB L-0501
Number analyzed (Participants) | 4
ng・h/mL | 9218.56 (6696.81)

16. Secondary Outcome: The Half-life Period (t1/2) of Unchanged SyB L-0501 in Korea
Time Frame: as for outcome 9
Measure: Median (Standard Deviation); unit: hour
Arm/Group | SyB L-0501
Number analyzed (Participants) | 4
hour | 0.48 (0.18)

ADVERSE EVENTS:
Time Frame: up to 30 weeks
Arm/Group | SyB L-0501
Serious Adverse Events (participants affected / at risk) | 14/59
Other Adverse Events (participants affected / at risk) | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SyB L-0501 (N=59)
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Death (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Cytomegalovirus infection (Infections and infestations) | 3
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Pneumonia cytomegaloviral (Infections and infestations) | 1
Gastric cancer (Infections and infestations) | 1
Urinary retention (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SyB L-0501 (N=59)
Anaemia (Blood and lymphatic system disorders) | 30
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 12
Lymphopenia (Blood and lymphatic system disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 16
Arrhythmia supraventricular (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Anal ulcer (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 29
Diarrhoea (Gastrointestinal disorders) | 8
Dysphagia (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 20
Oral discomfort (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Periodontitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 6
Epigastric discomfort (Gastrointestinal disorders) | 1
Oral mucosa erosion (Gastrointestinal disorders) | 1
Application site reaction (General disorders) | 1
Asthenia (General disorders) | 7
Chest discomfort (General disorders) | 1
Chills (General disorders) | 1
Face oedema (General disorders) | 2
Fatigue (General disorders) | 13
Feeling hot (General disorders) | 3
Generalised oedema (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection site erythema (General disorders) | 1
Injection site pain (General disorders) | 1
Injection site phlebitis (General disorders) | 1
Injection site reaction (General disorders) | 3
Malaise (General disorders) | 14
Mucosal inflammation (General disorders) | 4
Multi-organ failure (General disorders) | 1
Oedema (General disorders) | 4
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 15
Infusion site reaction (General disorders) | 1
Inflammation (General disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Liver injury (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 2
Gastrointestinal infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 4
Infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 4
Oral candidiasis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Enterocolitis infectious (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 4
Fall (Injury, poisoning and procedural complications) | 1
Tooth injury (Injury, poisoning and procedural complications) | 1
Open wound (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 19
Aspartate aminotransferase increased (Investigations) | 22
Blood albumin decreased (Investigations) | 1
Blood bilirubin increased (Investigations) | 2
Blood chloride increased (Investigations) | 1
Blood creatinine increased (Investigations) | 8
Blood immunoglobulin A decreased (Investigations) | 24
Blood immunoglobulin G decreased (Investigations) | 26
Blood lactate dehydrogenase increased (Investigations) | 20
Blood potassium increased (Investigations) | 2
Blood urea decreased (Investigations) | 4
Blood urea increased (Investigations) | 6
Blood uric acid decreased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
C-reactive protein increased (Investigations) | 23
CD4 lymphocytes decreased (Investigations) | 41
Eosinophil count increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 16
Glucose urine present (Investigations) | 3
Glycosylated haemoglobin increased (Investigations) | 1
Blood urine present (Investigations) | 1
Haemoglobin decreased (Investigations) | 2
Liver function test abnormal (Investigations) | 2
Lymphocyte count decreased (Investigations) | 33
Neutrophil count decreased (Investigations) | 34
Platelet count decreased (Investigations) | 26
Protein total decreased (Investigations) | 16
Red blood cell count decreased (Investigations) | 5
Weight decreased (Investigations) | 11
Weight increased (Investigations) | 4
White blood cell count decreased (Investigations) | 37
White blood cell count increased (Investigations) | 27
Blood bilirubin decreased (Investigations) | 1
Platelet count increased (Investigations) | 1
Basophil percentage increased (Investigations) | 1
Eosinophil percentage decreased (Investigations) | 1
Eosinophil percentage increased (Investigations) | 3
Monocyte percentage decreased (Investigations) | 2
Monocyte percentage increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 11
Hepatitis B virus test positive (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 7
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Hypouricaemia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Burning sensation (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 6
Headache (Nervous system disorders) | 10
Hypoaesthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 14
Major depression (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 10
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Photodermatosis (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 4
Phlebitis (Vascular disorders) | 1
Vasculitis (Vascular disorders) | 2
Haemorrhage (Vascular disorders) | 1
Angiopathy (Vascular disorders) | 3
Hot flush (Vascular disorders) | 5
Thirst (Gastrointestinal disorders) | 1
Blood immunoglobulin M decreased (Investigations) | 25
Neutrophil count increased (Investigations) | 22
Bone pain (Musculoskeletal and connective tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No